CLINICAL TRIAL: NCT05106049
Title: Early Detection of Renal Impairment in Patients With Non-alcoholic Fatty Liver Disease by Measuring Serum Adiponectin Level.
Brief Title: Serum Adiponectin as an Early Marker for Renal Impairment in Patients With Non-alcoholic Fatty Liver Disease.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hend Abdelrheem Ahmed, Hend Abdelrheem, Assiut University
Other Study IDs: Adiponectin in NAFLD
Record Dates: First submitted 2021-10-23; First posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases: non-alcoholic fatty liver patients
  Interventions: Diagnostic Test: serum Adiponectin
- control: healthy persons
  Interventions: Diagnostic Test: serum Adiponectin

INTERVENTIONS:
Diagnostic Test: serum Adiponectin — serum adiponectin as early marker for renal impairment. Adiponectin is a recently identified adipose tissue-derived protein (adipocytokine) with important metabolic ,antiinflammatory, anti-atherogenic, and reactive oxygen species protective actions.

SUMMARY:
Early detection of renal impairment in patients with non-alcoholic fatty liver disease and its correlation with serum Adiponectin level.

DETAILED DESCRIPTION:
Detection of serum Adiponectin by ELISA technique using (EIA-3418) KIT, DRG international inc., USA

ELIGIBILITY:
Inclusion Criteria:

* Patients with fatty liver aged from 18 to 60 yrs either diabetic or not .
* Patient with normal echogenic kidney in ultrasound and eGFR more than 60 mL/min/1.73m2.
* The Control group are completely healthy subjects without any systemic or liver and kidney affection

Exclusion Criteria:

* Patients less than 18 yrs & more than 60 yrs .
* All patients having any other causes of renal and hepatic disease rather than Diabetes and having any other systemic problem.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: cases are Non-alcoholic fatty liver patients who do not having any other health problem.
  control group is healthy individuals.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Correlate serum Adiponectin level with renal impairment in non-alcoholic fatty liver disease. | baseline
  measure level of serum Adiponectin in non-alcoholic fatty liver patients to detect early renal impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Hassan, Profissor.as, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stefan N, Stumvoll M. Adiponectin--its role in metabolism and beyond. Horm Metab Res. 2002 Sep;34(9):469-74. doi: 10.1055/s-2002-34785. PMID 12384822